CLINICAL TRIAL: NCT06687174
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Study to Evaluate the Efficacy and Safety of MY008211A in Subjects with Primary Immunoglobulin a Nephropathy (IgAN)
Brief Title: Study to Evaluate the Efficacy and Safety of MY008211A in Subjects with Primary Immunoglobulin a Nephropathy (IgAN)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wuhan Createrna Science and Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MY008211A-IgAN-2-01
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: IgA Nephropathy (IgAN)
Keywords: kidney disease; Primary glomerular disease
MeSH Terms: conditions — Glomerulonephritis, IGA; Kidney Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The trial was a double-blind design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MY008211A 200 mg BID (Experimental): 200 mg taken twice a day.
  Interventions: Drug: MY008211A tablets
- MY008211A 400 mg BID (Experimental): 400 mg taken twice a day.
  Interventions: Drug: MY008211A tablets
- Placebo (Placebo Comparator): Matching placebo to MY008211A taken twice a day.
  Interventions: Drug: MY008211A tablets matched placebo

INTERVENTIONS:
Drug: MY008211A tablets — MY008211A BID
  Arms: MY008211A 200 mg BID; MY008211A 400 mg BID
Drug: MY008211A tablets matched placebo — Matching placebo to MY008211A taken twice a day.
  Arms: Placebo

SUMMARY:
Efficacy and safety of MY008211A in IgAN patients

DETAILED DESCRIPTION:
This was a multicenter, randomized, double-blind, dose-ranging, parallel-group study. Two doses of MY008211A (200mg, 400mg) were compared with placebo. The study comprised a screening period of this study for 90 days, an efficacy observation period for 24 weeks, a long-term study for 80 weeks, and a follow-up period for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 18 and ≤ 75 years of age at Screening.
2. Estimated GFR(eGFR) ≥30 mL/min/1.73m2.
3. Subjects with a biopsy-confirmed diagnosis of IgAN.
4. Urine protein ≥0.75 g/24h from a 24h urine collection.
5. All patients must have been on stable supportive care including a maximally tolerated dose or approved maximal dose of ACEi or ARB therapy for at least 90 days prior to the first administration of study drug.
6. Subjects who received SGLT2i must have been on a stable treatment with the maximum allowed or tolerated dose prior to the first administration of study drug.
7. Vaccination against Neisseria meningitidis(MenACWY) is required within 3 years.
8. Vaccination for the prevention of S. pneumoniae is required within 5 years.

Exclusion Criteria:

1. Systolic blood pressure >130 mm Hg or diastolic blood pressure >80 mm Hg.
2. Presence of any secondary IgAN.
3. Presence of rapidly progressive glomerulonephritis.
4. Presence of other chronic kidney diseases.
5. Patients with a diagnosis of type 1 or type 2 diabetes mellitus.
6. A history of invasive infections caused by encapsulated bacteria, e.g., meningococci or pneumococci.
7. Patients previously treated with immunosuppressive agents exposure within 90 days prior to start of study drug dosing.
8. Patients previously treated with traditional Chinese medicine containing immunosuppressive ingredients within 90 days prior to start of study drug dosing.
9. Patients who had been treated with any systemic corticosteroids within the 180 days before treatment ≥20 mg/d for primary IgAN indication.
10. Patients who previously have received biologic agent or monoclonal antibodies prior to start of study drug dosing within 5 half-lives or 30 days (whichever is longer).
11. Patients who have received live/attenuated vaccines within the 4 weeks prior to randomization, or plan to receive during the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
The ratio of urine protein to creatinine concentration ratio (UPCR based on 24h urine collection, 24h-UPCR) relative to baseline at Week 12. | Week 12
  Participants collected their urine over a 24-hour period.

SECONDARY OUTCOMES:
The ratio of 24 h-UPCR relative to baseline at each visit during treatment period except Week 12. | up to 24 weeks
  Participants collected their urine over a 24-hour period.
The ratio of 24-hour urine protein excretion (24 h-UPE) relative to baseline at each visit during treatment period. | up to 24 weeks
  Participants collected all of their urine over a 24-hour period.
The ratio of 24-hour urine albumin (24 h-UA) relative to baseline at each visit during treatment period. | up to 24 weeks
  Participants collected all of their urine over a 24-hour period.
The ratio of 24-hour urine albumin to creatinine concentration ratio (24 h-UACR) relative to baseline at each visit during treatment period. | up to 24 weeks
  Participants collected all of their urine over a 24-hour period.
Change from baseline in serum creatinine at each visit during treatment period. | up to 24 weeks
  Serum creatinine
Change from baseline in estimated glomerular filtration rate (eGFR) at each visit during treatment period. | up to 24 weeks
  eGFR was calculated according to the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI).

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zhang, PH.D., Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China